CLINICAL TRIAL: NCT05631886
Title: A Pilot Clinical Trial of Autologous EphA-2-Targeting Chimeric Antigen Receptor Dendritic Cell Vaccine Loaded With TP53 Mutant Peptide Plus ICIs for Local Advanced/Metastatic Solid Tumors or Relapsed/Refractory Lymphomas.
Brief Title: Combination of CAR-DC Vaccine and ICIs in Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-075
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor, Adult; Lymphoma; EphA2 Overexpression; TP53 R273H; TP53 R175H; TP53 R248Q; TP53 R249S
Keywords: Local Advanced/Metastatic; Relapsed/refractory
MeSH Terms: conditions — Lymphoma; Neoplasm Metastasis; Recurrence | interventions — Albumin-Bound Paclitaxel; Cyclophosphamide; Injections; spartalizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TP53-EphA-2-CAR-DC plus anti-PD-1 antibody/anti-CTLA4 antibody (Experimental): In the priming phase, a conditioning chemotherapy regimen of Abraxane and cyclophosphamide is administered three days before vaccination, and TP53-EphA-2-CAR-DC vaccine is infused on Day 0 and Day 7 in Week 1.
  In the boost phase, TP53-EphA-2-CAR-DC vaccine is infused one dose every 8 weeks since Week 5.
  Anti-PD-1 antibody and anti-CTLA4 antibody are administered 2 days after the first dose of TP53-EphA-2-CAR-DC vaccine in the boost phase (Day 3 in Week 5) and every 3 weeks afterwards for four doses, followed by anti-PD-1 antibody once every 3 weeks, until:
  1. Unacceptable toxicity occurred or disease progression; or 2. Reactive T cells are undetected repeatedly after the last vaccine dose; or 3. Vaccine exhaustion.
  Interventions: Biological: TP53-EphA-2-CAR-DC; Drug: Abraxane; Drug: Cyclophosphamide; Drug: anti-PD-1 antibody; Drug: Anti-CTLA4 Monoclonal Antibody

INTERVENTIONS:
Biological: TP53-EphA-2-CAR-DC — 5~10 × 10^6 CAR DCs per dose will be administered by intravenous injection.
Drug: Abraxane — Intravenous abraxane 125 mg/m^2/day on day-5.
  Other Names: Abraxane Injectable Product
Drug: Cyclophosphamide — Intravenous cyclophosphamide 300 mg/m^2/day on day -4.
  Other Names: Cyclophosphamide for Injection
Drug: anti-PD-1 antibody — Intravenous anti-PD-1 antibody 200 mg/day.
  Other Names: PD-1 blocking antibody
Drug: Anti-CTLA4 Monoclonal Antibody — Intravenous anti-CTLA4 antibody 1 mg/kg/day
  Other Names: Ipilimumab

SUMMARY:
This is a pilot clinical trial for subjects with local advanced/metastatic solid tumors or relapsed/refractory (R/R) lymphomas to determine the safety, efficacy and immune response of autologous EphA2-targeting CAR-DC vaccine loaded with TP53 mutant peptide (TP53-EphA-2-CAR-DC) in combination with ICIs. It aims to: assess the safety and antitumor effects of TP53-EphA-2-CAR-DC vaccine; detect T cell response against TP53 mutant peptide and tumor neoepitopes after the treatment with TP53-EphA-2-CAR-DC vaccine and ICIs.

DETAILED DESCRIPTION:
Therapeutic cancer vaccines, especially DC-based vaccines, are extensively pursued immune approaches in addition to immune checkpoint blockade antibodies and chimeric antigen receptor T cells. DCs can engulf, process and present tumor antigens to T cells, thereby initiating a potent and tumor-specific immune response. However, clinical outcomes of therapeutic cancer vaccines still remain poor, with objective response rates that rarely exceed ~15%. The maturation and activation of DCs are necessary steps to trigger the antitumor responses. However, it is increasingly clear that tumor-infiltrating dendritic cells (TIDCs) usually have an immature or tolerated phenotype that plays central roles in developing tumor microenvironment (TME). As a consequence, malfunction of TIDCs could suppress the infiltration and function of tumor infiltrating T cells and convert them into immune suppressive regulatory T cells.

In our previous research, we constructed novel CAR-DCs (Chimeric antigen receptor engineered dendritic cells) containing a scFv domain targeting EphA2 antigen, CD8a transmembrane, tandem DC-specific activation domains. The engineered CAR-DCs were activated when contacting with tumor targets in TME, and consequently, augmented the cytotoxicity of antigen specific T cells in immune system humanized solid tumor mouse models. Our design of CAR-DCs provides an effective vaccine strategy for malignant tumors. Therefore, we designed an autologous CAR-DC vaccine engineered with anti-EphA2 CAR and TP53 mutant peptide (TP53-EphA-2-CAR-DC), which can suppress the growth of tumors expressing the correlated TP53 mutant in animal models. In addition, the combination of the immune checkpoint inhibitors could further reverse immunosuppressive TME and globally activate T cell responses. In this pilot study, we aim to assess the safety, efficacy and immune response of TP53-EphA-2-CAR-DC combined with anti-PD-1 antibody/anti-CTLA4 antibody in patients with local advanced/metastatic solid tumors or R/R lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (inclusive).
2. ECOG performance status ≤2 and Estimated life expectancy of more than 3 months.
3. Local advanced/metastatic solid tumors or R/R lymphomas confirmed by histopathology or cytology with documentation of tumor EphA2 positive (≥20%) and TP53 mutation (R273H or R175H or R248Q or R249S) within 6 months prior to screening. The second malignancy is allowed.
4. No clinical response to standard frontline therapy or no standard therapy exists for solid tumors. Relapse after treatment with ≥2 lines systemic therapy or refractory disease for lymphomas. Patients who have declined standard therapy or have no access to standard therapy may be enrolled and the reasons for a lack of access need to be documented. Previous treatment with anti-PD-1/PD-L1 antibodies or anti-CTLA4 antibody are allowed, regardless of the level of PD-1/PD-L1 expression, dMMR and TMB.
5. At least one measurable lesion at baseline per RECIST version 1.1 or Lugano response criteria 2014.
6. Adequate organ function as defined by the following criteria: ANC ≥1000 cells/μL; Platelet count ≥80,000/μL; Hemoglobin ≥8.0 g/dL (hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions); Serum AST and serum ALT, ≤3.0 x ULN (≤5 x ULN for patients with liver metastases); Total serum bilirubin ≤3.0 x ULN); Serum creatinine ≤2 x ULN or creatinine clearance of ≥45 mL/min.
7. Willing to undergo either excised or large-needle lymph node or tissue biopsy, or provide formalin-fixed paraffin-embedded (FFPE) tumor tissue block or freshly cut unstained slides.
8. Willing to complete all scheduled visits and assessments at the institution administering the therapy.
9. Able to read, understand and provide written informed consent.

Exclusion Criteria:

1. Having TP53 (R273H or R175H or R248Q or R249S) germline mutation.
2. Active central nervous system disease involvement (but allow patients with prior brain metastases treated at least 4 weeks prior to enrollment that are clinically stable and do not require intervention), or prior history of NCI CTCAE Grade ≥3 drug-related CNS toxicity.
3. Prior organ allograft transplantations or allogeneic hematopoietic stem cell transplantation.
4. Evidence of active uncontrolled viral, bacterial, or systemic fungal infection.
5. Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS).
6. Active infection of hepatitis B virus (HBV), or hepatitis C virus (HCV).
7. Patients with history (within the last 5 years) or risk of autoimmune disease who have immunosuppressive medications or immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone or equivalent) within 28 days prior to enrollment. However, patients who received a short course of corticosteroids (eg, premedication prior to antibody drug) will be eligible for study entry.
8. Major trauma or major surgery within 4 weeks prior to enrollment.
9. Previous treatment involving TP53 mutant (R273H or R175H or R248Q or R249S) and EphA2.
10. Systemic chemotherapy and other intervene within 2 weeks prior to vaccination.
11. Being participating or withdrew any other trials within 4 weeks.
12. Any serious underlying medical (eg, pulmonary, renal, hepatic, gastrointestinal, or neurological) or psychiatric condition or any issue that would limit compliance with study requirements.
13. Vaccination within 30 days of study enrollment.
14. Pregnant, lactating, or breastfeeding females.
15. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events (AEs) | 2 years
  Determining the safety profile following the initiation of treatment and grading these toxicities by CTCAE v5.0. AEs such as cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Clinical Response | 2 years
  Clinical Response will be determined by iRECIST criteria. Response rate is the proportion of patients that achieve CR or PR.
Immune Response | Peripheral blood: baseline, weekly before Week 9, prior to each vaccination after Week 9 until last vaccine and 1 year after last vaccine. Tumor tissue: baseline, Week 3, and following timing will be performed according to subject's condition.
  Immune response will be evaluated by phenotype and functional analysis of vaccine-reactive T cells and Neoantigen-reactive T cells as well as other immune cells in peripheral blood and tumor samples. Response is defined by ≥3 folds increase relative to pre-vaccination.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  PFS is defined as the time from TP53-EphA-2-CAR-DCs infusion to documented disease progression or death.
Overall Survival (OS) | 2 years
  OS is defined as the time from TP53-EphA-2-CAR-DCs infusion to the date of death.
Time to response (TTR) | 2 years
  TTR is defined as the time from TP53-EphA-2-CAR-DCs infusion to first assessed CR or PR by investigators and based on the iRECIST criteria.
Duration of response (DOR) | 2 years
  DOR is defined as the time from objective response (OR) until documented tumor progression date among responders.
Number and copy number of TP53-EphA-2-CAR-DCs | Peripheral blood samples are collected on days 0, 3, 7, 10, 22, the day before each vaccination until last vaccination and 1 year after last vaccine. Tumor tissues are collected at baseline, the day before Week 5, and after combination.
  Number and copy number of TP53-EphA-2-CAR-DCs were assessed by the number in peripheral blood and tumor tissue.
The level of cytokines in serum | Peripheral blood samples are collected on days 0, 3, 7, 10, 22, the days before each vaccination until last vaccination and 1 year after last vaccine. Tumor tissues are collected at baseline, the day before Week 5, and after combination.
  The cytokines mainly include IL-1, IL-2, IL-6, IL-8, IL-10, IL-12 (p70), TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xu, Ph.D, Study Director — Zhejiang University
Locations (1):
- Biotherapeutic Department of Chinsese PLA Gereral Hospital, Beijing, Beijing Municipality, China